CLINICAL TRIAL: NCT02119078
Title: Acute Care for Elders (ACE) Program at OHSU Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Juliana Bernstein, Assistant Professor, Physician Assistant, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RB00010420
Record Dates: First submitted 2014-04-08; First posted 2014-04-21 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Delirium; Age-Related Cognitive Decline; Frail Elderly; Hospital Acquired Pressure Ulcer; Drug-Related Side Effects and Adverse Reactions
Keywords: Geriatrics; Acute Care for Elders; Geriatric syndromes; Delirium; Falls; Polypharmacy
MeSH Terms: conditions — Delirium; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE Service (Active Comparator): Admission to the Acute Care for Elders (General Medicine Team 1) service. (See Intervention, below)
  Interventions: Other: Acute Care of Elders focused geriatric care
- Standard care (other General Medicine teams) (No Intervention): Admission to one of the 4 non-ACE general medicine teaching teams at OHSU.

INTERVENTIONS:
Other: Acute Care of Elders focused geriatric care — Patients admitted to the ACE Service will receive standard care as well as additional use of geriatric-specific order sets and protocols and oversight of care by a geriatric-trained Advanced Practice Provider (APP).
  Arms: ACE Service

SUMMARY:
The purpose of this investigation is to assess the effectiveness of a multi-disciplinary Acute Care for Elders (ACE) program dedicated to the care of patients age 70 and older admitted to Oregon Health & Science University's hospital medicine service. The ACE program will aim to improve the quality of care of older patients in the investigators hospital by implementing focused interventions and recommendations specific to geriatric needs and syndromes, including: reduced fall rate, decreased incidence and duration of delirium, early recognition and treatment of impaired mobility and function, careful minimization of medication use, prevention of unnecessary catheter and restraint use, decreased hospital readmission rates, improved transitional care following hospital discharge, and high levels of patient and referring physician satisfaction. Additionally, the ACE program aims to improve resident and student competence in treating geriatric syndromes, and to improve staff and learner satisfaction with caring for older adults. ACE programs have been well studied at other institutions, so the investigators will be implementing a program that is already standard of care, and studying the elements that are unique to OHSU.

This will be a quality improvement project. Study participants will be a convenience sample of OHSU faculty, staff, residents and students who are employed by or on rotation with General Medicine Team 1 of the Medicine Teaching Service. Faculty, staff, and learners (ACE team members) will receive the ACE training. Study personnel will conduct prospective and retrospective chart review of patients admitted to the ACE service to determine outcomes as noted above.

ELIGIBILITY:
Inclusion Criteria (ACE faculty, health care providers and students):

* employed by OHSU or enrolled in one of OHSU's schools (medicine, nursing, pharmacy)
* share in the care of older adults on the General Medicine Team 1 service.

Inclusion Criteria (patients):

* admitted to the internal medicine service during the time frame of the study
* age 70 or older at time of hospital admission

Exclusion Criteria (ACE faculty, health care providers and students):

* non-English-speaking

Exclusion Criteria (patients):

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-06-30 (Actual); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of geriatric patients with adverse events | During hospitalization, an expected average of 6 days
  Incidence and duration of delirium (source: hospital problem list); incidence of hospital-acquired pressure ulcers (source: nursing documentation, problem list); number of prescriptions for Beers List medications during hospitalization and upon discharge (source: MAR)

SECONDARY OUTCOMES:
Resident confidence in treating geriatric syndromes | After 3 week rotation on the Acute Care for Elders service
  As measured by the Post-ACE Survey resident questionnaire, which includes 17 metrics of confidence (e.g. management of pain, identification of fall risk factors, delivering bad news, discussion of hospice care, performing a complete skin exam, documenting advanced directives, managing insomnia, performing bedside cognitive assessments.)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana M Bernstein, MPAS, PA-C, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University Hospital, Portland, Oregon, United States